CLINICAL TRIAL: NCT05431556
Title: Pilot Study of Virtual Mind-Body Exercises for Patients Undergoing Pancreatic Surgery
Brief Title: Virtual Mind-Body Exercises for People Having Pancreatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-070
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Pancreas Disease
Keywords: Exercises; 22-070
MeSH Terms: conditions — Pancreatic Diseases; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual mind-body group exercise classes (VMB) (Experimental): Will be provided with the schedule and links to the web-based mind-body exercises offered by MSK in real-time via the Zoom video conferencing platform. Each session is led by a licensed clinician (e.g., licensed dance therapist, certified yoga instructor, nurse specialist/physical trainer) with specific expertise in the oncology setting.
  Interventions: Other: Virtual mind-body group exercise classes
- Enhanced usual care (EUC) (Active Comparator): Pre-recorded self-care videos.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Other: Virtual mind-body group exercise classes — Pre-operative period (baseline/intake day to day before surgery): mid- to high intensity classes focusing on aerobic physical activity, relaxation, and stress management (classes: Fitness for Everyone, Tai Chi, Mat Yoga, Dance Cardio, Meditation, Core Strength, Music Therapy)
  * Immediate post-operative period (post-operative hospitalization to 2 weeks after surgery): low- to mid-intensity classes focusing on relaxation, stress management and low-impact physical activity (classes: Chair Yoga, Dance Therapy, Meditation, Music Therapy)
  * Late post-operative period (3-12 weeks after surgery): mid- to high-intensity classes focusing on aerobic physical activity, relaxation, and stress management (classes: Fitness for Everyone, Tai Chi, Mat Yoga, Dance Cardio, Meditation, Core Strength, Music Therapy)
  Arms: Virtual mind-body group exercise classes (VMB)
Other: Enhanced usual care — EUC arm will be referred to MSK's multimedia page on the Integrative Medicine website to access pre-recorded mind-body videos on their own time. These videos are 15-60 minutes in duration and consist of educational and self-care videos, including guided meditation and Tai Chi.
  Arms: Enhanced usual care (EUC)

SUMMARY:
The purpose of this study is to find out if it is practical to provide 2 interventions, VMB exercise classes and EUC (pre-recorded self-care videos), during the perioperative period (before and after surgery) to improve health-related outcomes and quality of life for people undergoing a pancreatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older
* Any pancreas disease (benign, pre-malignant, or malignant) and will be undergoing pancreatectomy
* Has at least one week to participate in the study prior to the anticipated surgery date
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1
* English-speaking only

Exclusion Criteria:

* Unable to give informed consent due to cognitive impairment or impaired decisionmaking capacity
* Cognitive impairment precluding response to study assessments
* Received neoadjuvant or any chemoradiation in the past 60 days
* Unwilling to accept random assignment
* Unwilling to commit to the 12-week study time period
* Unlikely to be compliant because of social factors that prevent patients from attending classes or doing home practice (e.g., unreliable internet, no access to a computer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Virtual Mind-Body Exercises program as measured by enrollment rate | 1 year
  total number of patients invited, and the total number of study participants will be recorded

SECONDARY OUTCOMES:
improving patient-reported outcomes (PROs) | 1 year
  Changes in HADS anxiety scores. The Hospital Anxiety and Depression Scale (HADS) will be used to explore the effect of treatments on psychological distress, specifically on anxiety. HADS is a 14-item scale with seven items measuring depression and seven items measuring anxiety. Each item is answered by the patient on a four-point (0-3) response category; possible scores range from 0-21 for anxiety and depression, with higher scores indicating higher symptomatology. Established cutoffs are: 0-7 not significant; 8-10 subclinical; and 11-21 clinically significant depression/anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Wei, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm